CLINICAL TRIAL: NCT03057977
Title: A Phase III Randomised, Double-blind Trial to Evaluate Efficacy and Safety of Once Daily Empagliflozin 10 mg Compared to Placebo, in Patients With Chronic Heart Failure With Reduced Ejection Fraction (HFrEF)
Brief Title: EMPagliflozin outcomE tRial in Patients With chrOnic heaRt Failure With Reduced Ejection Fraction (EMPEROR-Reduced)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.121; 2016-002280-34 (EudraCT Number)
Record Dates: First submitted 2017-02-16; First posted 2017-02-20 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — once daily
  Other Names: JARDIANCE, JARDIANZ, GIBTULIO
  Arms: Empagliflozin
Drug: Placebo — once daily
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate the safety and efficacy of empagliflozin versus placebo on top of guideline-directed medical therapy in patients with heart failure with reduced ejection fraction.

ELIGIBILITY:
Inclusion criteria:

* Male or female patient age >= 18 years at screening. For Japan only: Age >= 20 years at screening
* Patients with chronic HF (Chronic Heart Failure) NYHA (New York Heart Association Classification) class II-IV and reduced EF (Ejection Fraction) (LVEF (Left Ventricular Ejection Fraction) <=40%) and elevated NT-proBNP (N-terminal of the prohormone brain natriuretic peptide)

  * If EF >= 36% to <= 40%: NT-proBNP >= 2500 pg/ml or patients without AF (atrial fibrillation/atrial flutter) and NT-proBNP >= 5000 pg/ml for patients with AF
  * If EF >= 31% to <= 35%: NT-proBNP >= 1000 pg/ml for patients without AF and NT-proBNP >=2000 pg/ml for patients with AF
  * If EF<= 30%: NT-proBNP >= 600 pg/ml for patients without AF and NT-proBNP >=1200 pg/ml for patients with AF
  * EF ≤ 40% and hospitalization for heart failure in the past 12 months: NTproBNP ≥ 600 pg/ml for patients without AF and NT-proBNP >= 1200 pg/ml for patients with AF
* Appropriate dose of medical therapy for HF consistent with prevailing local and international CV (Cardiovascular) guidelines, stable for at least 1 week prior to Visit 1
* Appropriate use of medical devices such as cardioverter defibrillator (ICD) or a cardiac resynchronization therapy (CRT) consistent with prevailing local or international CV guidelines
* Signed and dated written ICF (Informed Consent Form)
* Further inclusion criteria apply

Exclusion criteria:

* Myocardial infarction, coronary artery bypass graft surgery, or other major cardiovascular surgery, stroke or TIA (Transient Ischaemic Attack) in past 90 days prior to Visit 1
* Heart transplant recipient, or listed for heart transplant
* Acute decompensated HF
* Systolic blood pressure (SBP) >= 180 mmHg at Visit 2.
* Symptomatic hypotension and/or a SBP < 100 mmHg
* Indication of liver disease
* Impaired renal function, defined as eGFR (Estimated Glomerular Filtration Rate) < 20 mL/min/1.73 m2 (CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration Equation)) or requiring dialysis
* History of ketoacidosis
* Current use or prior use of a SGLT (Sodium-glucose co-transporter)-2 inhibitor or combined SGLT-1 and 2 inhibitor
* Currently enrolled in another investigational device or drug study
* Known allergy or hypersensitivity to empagliflozin or other SGLT-2 inhibitors
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3730 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (519):
- United States (92):
  - La Mesa Cardiac Center, La Mesa, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Merced Vein and Vascular Center, Merced, California
  - University of California Irvine, Orange, California
  - Covigilant Research, LLC, Riverside, California
  - University of California, Torrance, California
  - Orange County Research Center, Tustin, California
  - Blue Coast Cardiology, Vista, California
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Integrated Heart Care, Boca Raton, Florida
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Integrative Research Associates, Fort Lauderdale, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Cardiology Consultants, Inc, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Grady Clinical Research Center, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Cardiovascular Group PC, Lawrenceville, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - University of Chicago, Chicago, Illinois
  - Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Rockford Cardiovascular Associates, Rockford, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - St. Francis Medical Group-Indiana Heart Physicians, Inc, Indianapolis, Indiana
  - Reid Hospital, Richmond, Indiana
  - Beacon Medical Group Clinical Research, South Bend, Indiana
  - Research Integrity, LLC, Owensboro, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Louisiana Heart Center, Covington, Louisiana
  - Clinical Trials of America, LLC, Monroe, Louisiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins University Hospital School of Medicine, Baltimore, Maryland
  - MedStar Health Research Institute, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants, Beltsville, Maryland
  - Spectrum Clinical Research, Towson, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - East Mountain Medical Associates, PC, Great Barrington, Massachusetts
  - Alpena General Hospital, Alpena, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Louis University, St Louis, Missouri
  - SLHV, St Louis, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Trinity Medical WNY, PC, Cheektowaga, New York
  - Northwell Health, Great Neck, New York
  - Mount Sinai School of Medicine, Lake Success, New York
  - St. Luke's Roosevelt Hospital, New York, New York
  - Harlem Cardiology, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Cardiac Care and Vascular Medicine, PLLC, The Bronx, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Kernodle Clinic West, Burlington, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Clinical Trials of America, Inc, Lenoir, North Carolina
  - Rama Research LLC, Marion, Ohio
  - University of Toledo, Toledo, Ohio
  - South Oklahoma Heart Research Group, Oklahoma City, Oklahoma
  - Doylestown Health Cardiology, Doylestown, Pennsylvania
  - York Hospital, WellSpan Health, York, Pennsylvania
  - AnMed Health Clinical Research, Anderson, South Carolina
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Palmetto Health, Columbia, South Carolina
  - William Jennings Bryan Dorn VA Medical Center, Columbia, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Palmetto Research Center, LLC, Spartanburg, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Soltero Cardiovascular Research Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of North Texas Health Science Center, Fort Worth, Texas
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital, Plano, Texas
  - Alpine Research Organization, Farmington, Utah
  - Cardiac Health Management Network, P.C., Chester, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Roanoke Heart Institute PLC, Roanoke, Virginia
  - Salem VA Medical Center, Salem, Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
- Argentina (40):
  - Hospital Interzonal General de Agudos Dr Jose Penna, Bahía Blanca
  - Hospital Italiano Regional del Sur, Bahia Blanca, Bahía Blanca
  - CIPREC, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Consultorios Asociados de Endocrinología e Invest Clínica, Ciudad Autonoma Buenos Aires
  - Instituto Cardiovascular de Buenos Aires, Ciudad Autonoma Buenos Aires
  - CCBR - Buenos Aires - AR, Ciudad Autonoma Buenos Aires
  - Centro Médico Viamonte, Ciudad Autonoma de Bs As
  - Sanatorio Güemes, Ciudad Autónoma de Bs As
  - Instituto Medico Elsa Perez SRL (IMEP), Ciudadela
  - Clinica Coronel Suarez SA, Coronel Suárez
  - Instituto de Cardiología de Corrientes, Corrientes
  - Sanatorio Mayo Privado SA, Córdoba
  - Centro de Investigaciones Clinicas Instituto del Corazon, Córdoba
  - Sanatorio Allende S.A., Córdoba
  - Clínica Colombo, Córdoba
  - Instituto Médico DAMIC S.R.L., Córdoba
  - Hospital Privado, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Centro de Investigaciones Médicas, Mar del Plata
  - Hospital Privado de Comunidad, Mar del Plata
  - Clínica Olivos, Olivos
  - CER Instituto Médico, Quilmes
  - Instituto de Investigaciones Clínicas de Quilmes, Quilmes
  - Instituto de Investigaciones Clinicas de Rosario, Rosario
  - Instituto Medico Fundación Grupo Colaborativo Rosario, Rosario
  - Sanatorio Británico, Rosario
  - Sanatorio Plaza, Rosario
  - Sanatorio Parque, Rosario
  - Instituto CAICI, Rosario
  - CORDIS S.A., Salta, Salta
  - Centro Cardiovascular Salta, Salta
  - Corporacion Medica de Gral. San Martin S.A., San Martín
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán
  - Instituto de Cardiología, San Miguel de Tucumán
  - CCBR Tucuman, San Miguel de Tucumán
  - Centro Medico Luquez, San Vicente
  - Centro de Investigaciones Clínicas del Litoral, Santa Fe
  - Hospital "Dr. José Maria Cullen ", Santa Fé
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro
- Australia (9):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - CORE Research Group, Milton, Queensland
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - SA-Heart Ashford Specialist Centre, Ashford, South Australia
  - Heart and Vascular Research, Fullarton, South Australia
  - The Northern Hospital, Epping, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - University Hospital Geelong, Geelong, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (10):
  - AZ Sint-Jan Brugge, Bruges
  - C.H.U. de Charleroi, Charleroi
  - AZ Sint-Blasius, Dendermonde
  - Ziekenhuis Oost-Limburg - Campus Sint-Jan, Genk
  - AZ Sint-Lucas - Campus Sint Lucas, Ghent
  - Grand Hôpital de Charleroi, Gilly
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - La Louvière - UNIV CHU Tivoli, La Louvière
  - UZ Leuven, Leuven
  - AZ Sint-Maarten, Mechelen
- Brazil (38):
  - Hospital Felicio Rocho, Belo Horizonte
  - Hospital Vera Cruz, Belo Horizonte
  - Cardresearch Cardiologia Assistencial e de Pesquisas Ltda, Belo Horizonte
  - CCBR - Brasília, Brasília
  - ICDF - Instituto de Cardiologia do Distrito Federal, Brasília
  - CECAP - Centro de Cardiologia Clínica, Brasília
  - Hospital Angelina Caron, Campina Grande do Sul
  - Centro Especializado em Cardiol Loema Instituto de Pesq Clin, Campinas
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - CAEP - Centro Avançado de Estudos e Pesquisas Ltda.,Campinas, Campinas
  - Hospital Universitário, Canoas
  - IPCEM - Instituto de Pesquisa Clínica para Estudos Multicêntricos - Universidade de Caxias do Sul, Caxias do Sul
  - Irmandade da Santa Casa de Misericórdia de Curitiba, Curitiba
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes, Fortaleza
  - Barroso e Sebba Ltda, Goiânia
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - ICM - Instituto do Coracao de Marilia, Marília
  - Hospital São Vicente de Paulo, Passo Fundo
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Centro de Pesquisas em Diabetes, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Instituto de Cardiologia Rio Grande do Sul, Porto Alegre
  - Hospital Agamenon Magalhaes, Recife
  - H.C.da Fac. de Medicina de Ribeirao Preto, Ribeirão Preto
  - CCBR - Rio de Janeiro - BR, Rio de Janeiro
  - Hospital Universitário Pedro Ernesto UERJ, Rio de Janeiro - RJ
  - Pesquisare, Santo André
  - Praxis Pesquisa Médica, Santo André
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Fundacao Faculdade Regional de Medicina, Sao Jose, São José do Rio Preto
  - Centro de Pesquisa Clinica - CPCLIN, São Paulo
  - FGM - Clínica Paulista de Doenças Cardiovasculares, São Paulo
  - CDEC BRASIL - Centro de Desenvolvimento em Estudos Clínicos Brasil, São Paulo
  - Dr. Consulta, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica, São Paulo
  - INCOR e Hospital das Clínicas da Universidade de São Paulo, São Paulo
  - CEDOES - Diagnóstico e Pesquisa,Vitória, Vitória
  - Santa Casa de Votuporanga, Votuporanga
- Canada (30):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - G.A. Research Associates Ltd, Moncton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Brampton Cardio Pulmonary Clinic, Brampton, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - Cambridge Cardiac Care Inc., Cambridge, Ontario
  - Health Sciences North, Greater Sudbury, Ontario
  - Curnew Medicine Professional Corporation, Hamilton, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - M Heffernan Medicine Professional Corp., Oakville, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Heart Health Institute, Scarborough Village, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - North York Diagnostic and Cardiac Centre, Toronto, Ontario
  - Diabetes Heart Research Centre, Toronto, Ontario
  - Mohan Babapulle Medicine Professional Medicine, Waterloo, Ontario
  - Dr. Louis C.H. Yao, York, Ontario
  - ViaCar Recherche Clinique Inc, Greenfield Park, Quebec
  - Centre de Dépistage et Recherche Cardiovasculaire Rive-Sud, Longeuil, Quebec
  - Clinique Santé Cardio MC, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Centre de sante et de services sociaux de Beauce, Saint George-de-Beauce, Quebec
  - IUCPQ (Laval University), Québec
- China (27):
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - First Hospital of Jilin University, Changchun
  - Hunan Provincial People's Hospital, Changsha
  - 2nd Xiangya Hospital of Central South University, Changsha
  - The Third Hospital of Changsha, Changsha
  - Dongguan People's Hospital, Dongguan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Afiliated Hospital, Sun Yet-sen University, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Haikou People's Hospital, Haikou
  - HaiNan Provincial People's Hospital, Haikou
  - The First Affiliated Hospital of Lanzhou University, Lanzhou
  - The Second Affiliated Hospital of Lanzhou Medical University, Lanzhou
  - The Affiliated Hospital of Southwest Medical University, Luzhou
  - Nanchang University Affiliated 3rd Hospital, Nanchang
  - First Hospital Affiliated with Nanjing Medical University, Nanjing
  - Huashan Hospital, Fudan University, Shanghai
  - General Hospital of Shenyang Military Region, Shenyang
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Union Medical Center Nankai University Affiliated Hospital, Tianjin
  - Tongji Hospital, Tongji University, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Yanbian University Hospital, Yanji
  - the first people hospital of Yue Yang, Yueyang
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- Czechia (21):
  - Poliklinika Humanitas, Bílovec
  - Medicus Services Ltd., Brandys Nad
  - Internal and Cardiology Practice, MUDr. Karel Kamenik, Brno, Brno
  - MUDr. Alexandra Ludkova, Brno
  - Vojenska nemocnice Brno, Brno
  - Nemocnice Milosrdnych bratri, Brno
  - Edumed s.r.o, Broumov
  - MUDr. Jan Hubac, s.r.o. Kardiologicka ambulance, Chrudim
  - Nemocnice ve Frydku-Mistku, prispevkova organizace, Frýdek-Místek
  - MUDr. Ladislav Busak, Louny
  - Zdenek Vomacka, Olomouc
  - PV-Kardiologie s.r.o., Pardubice
  - General Faculty Hospital, Prague, Prague
  - University Hospital Motol, Prague
  - Thomayer Hospital, Praha 4 - Krc
  - Kardio Vaclavik s.r.o., Přerov
  - Clinic of Cardiology, Pribram, Příbram
  - Hospital Trebic, p.o., Třebíč
  - Masaryk Hospital, Usti nad Labem, Ústí nad Labem
  - Angiocor s.r.o, Zlín
  - KIGE s.r.o, Znojmo
- France (10):
  - HOP de Bayonne, Bayonne
  - HOP Jean Minjoz, Besançon
  - HOP Louis Pradel, Bron
  - HOP Côte de Nacre, Caen
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP La Pitié Salpêtrière, Paris
  - Centre Hospitalier de Pau, Pau
  - HOP Haut-Lévêque, Pessac
  - HOP Rangueil, Toulouse
  - INS Louis Mathieu, Vandœuvre-lès-Nancy
- Germany (31):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Praxis Dr. Rieker, Berlin, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Klinikum Bielefeld gGmbH, Bielefeld
  - Praxis Dr. Menzel, Dessau
  - St. Johannes Hospital Dortmund, Dortmund
  - Städtisches Klinikum Dresden, Dresden
  - GWT-TUD GmbH, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Studienzentrum Bocholderstraße, Essen
  - ClinPhenomics GmbH & Co KG, Frankfurt, Frankfurt
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen
  - Märkische Gesundheitsholding GmbH & Co. KG, Klinikum Lüdenscheid, Lüdenscheid
  - Praxis Dr. Sarnighausen, Lüneburg, Lüneburg
  - Katholisches Klinikum St. Hildegardiskrankenhaus, Mainz, Mainz
  - Deutsches Herzzentrum München, München
  - Kardiologische Gemeinschaftspraxis Nienburg, Nienburg
  - Kardiologische Praxis Papenburg, Papenburg
  - Universitätsklinikum Regensburg, Regensburg
  - Praxis Dr. Stenzel, Riesa, Riesa
  - Zentrum für Klinische Forschung, Wangen
  - Josephs-Hospital Warendorf, Warendorf
  - Petrus-Krankenhaus, Wuppertal
- Hungary (17):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Belgyogyaszati es Kardiologiai Maganrendelo, Békéscsaba
  - Clinexpert Kft., Budapest
  - Gottsegen Gyorgy Hungarian Instit.of Cardiology,Budapest, Budapest
  - Bajcsy-Zsilinszky Hospital and Clinic, Budapest
  - Semmelweis University, Budapest
  - Milit.Hosp.-State Health Cent., Budapest
  - Uzsoki Street Hospital, Budapest, Budapest
  - Nehezlegzes Ambulancia, Debrecen
  - Bugat Pal Hospital, Gyongyos, Gyöngyös
  - Selye Janos Hospital Komarom, Komárom
  - Dorottya Kanizsai Hospital, Nagykanizsa
  - Dr. Nagy Laszlo Kardiologiai Maganrendeles, Orosháza
  - Pecsi Tudomanyegyetem, Pécs
  - Da Vinci Maganklinika, Pécs
  - Fejer County Saint George University Teaching Hospital, Székesfehérvár
  - Veszpremi Sziv es Egeszseg Centrum, Veszprém
- India (14):
  - Doctor Jivraj Mehta Smarak Health Foundation, Ahmedabad
  - Kamalnayan Bajaj Hospital, Aurangabad
  - Narayana Institute of Cardiac Sciences, Bangalore
  - Rajarajeswari Medical College, Bengaluru
  - Madras Medical Mission,, Chennai
  - Apollo Speciality Hospital, Chennai
  - Medanta-The Medicity, Gūrgaon
  - B.M. Birla Heart research Centre, Kolkata
  - Vijan Cardiac and Critical Care Centre, Nashik
  - Siddhi Hospital, Nashik
  - Batra Hospital and Medical Research Centre, New Delhi
  - GB Pant Hospital, New Delhi
  - Fortis Escorts Heart Institute, New Delhi
  - Sir Gangaram Hospital, New Delhi
- Italy (10):
  - Azienda Ospedaliera G. Rummo, Benevento
  - ASST Papa Giovanni XXIII - A.O. Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Cona (FE)
  - Ospedale della Val di Chiana Santa Margherita, Cortona (AR)
  - Centro Cardiologico Monzino-IRCCS, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Umberto I Pol. di Roma-Università di Roma La Sapienza, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Azienda Servizi Sanitari 1 Triestina, Trieste
- Japan (66):
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Nagoya Kyoritsu Hospital, Aichi, Nagoya
  - Japanese Red Cross Nagoya Daini Hospital, Aichi, Nagoya
  - Toyota Memorial Hospital, Aichi, Toyota
  - Chiba Heart Clinic, Chiba, Chiba
  - Kimitsu Chuo Hospital, Chiba, Kisarazu
  - Seikeikai New Tokyo Heart Clinic, Chiba, Matsudo
  - Ehime Prefectural Central Hospital, Ehime, Matsuyama
  - Matsuyama Shimin Hospital, Ehime, Matsuyama
  - Uwajima City Hospital, Ehime, Uwajima
  - Fukuiken Saiseikai Hospital, Fukui, Fukui
  - Fukuoka University Chikushi Hospital, Fukuoka, Chikushino
  - Fukuokaken Saiseikai Futsukaichi Hospital, Fukuoka, Chikushino
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Aso Co.,Ltd Iizuka Hospital, Fukuoka, Iizuka
  - Steel Memorial Yawata Hospital, Fukuoka, Kitakyushu
  - Japan Community Health Care Organization Kyushu Hospital, Fukuoka, Kitakyushu
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - Chuno Kosei Hospital, Gifu, Seki
  - Fukuyama City Hospital, Hiroshima, Fukuyama
  - JA Hiroshima General Hospital, Hiroshima, Hatsukaichi
  - Shobara Red Cross Hospital, Hiroshima, Shobara
  - National Hospital Organization Hakodate Hospital, Hokkaido, Hakodate
  - Teine Keijinkai Clinic, Hokkaido, Sapporo
  - Tomakomai City Hospital, Hokkaido, Tomakomai
  - Hyogo Prefectural Amagasaki General Medical Center, Hyogo, Amagasaki
  - Hyogo Brain and Heart Center, Hyogo, Himeji
  - National Hospital Organization Kobe Medical Center, Hyogo, Kobe
  - Mito Medical Center, Ibaraki, Higashiibaraki-gun
  - National Hospital Organization Kanazawa Medical Center, Ishikawa, Kanazawa
  - Mitoyo General Hospital, Kagawa, Kanonji
  - Kagawa Prefectural Central Hospital, Kagawa, Takamatsu
  - Yamamoto Clinic, Kanagawa, Sagamihara
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Seiwakai Suizenji Touya Hospital, Kumamoto, Kumamoto
  - Kumamoto Rosai Hospital, Kumamoto, Yatsushiro
  - Uji-Tokushukai Medical Center, Kyoto, Uji
  - Sendai Kousei Hospital, Miyagi, Sendai
  - Sendai Tokushukai Hospital, Miyagi, Sendai
  - The Cardiovascular Center of Sendai, Miyagi, Sendai
  - National Hospital Organization Sendai Medical Center, Miyagi, Sendai
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Hokushin General Hospital, Nagano, Nakano
  - Nagasaki Medical Center, Nagasaki, Omura
  - Okayama City General Medical Center, Okayama, Okayama
  - Naha City Hospital, Okinawa, Naha
  - Nanbu Tokushukai Hospital, Okinawa, Shimajiri-gun
  - Urasoe General Hospital, Okinawa, Urasoe
  - Higashiosaka City Medical Center, Osaka, Higashiosaka
  - Kitano Hospital, Osaka, Osaka
  - Yodogawa Christian Hospital, Osaka, Osaka
  - Seichokai Bell Land General Hospital, Osaka, Sakai
  - Hokusetsu General Hospital, Osaka, Takatsuki
  - San-Ai Hospital, Saitama, Saitama
  - Kosekai Iwatsuki-minami Hospital, Saitama, Saitama
  - Kusatsu General Hospital, Shiga, Kusatsu
  - Tokushima Prefectural Central Hospital, Tokushima, Tokushima
  - National Hospital Organization Tokyo Medical Center, Tokyo, Meguro-ku
  - Ome Municipal General Hospital, Tokyo, Ome
  - Tokyo Rosai Hospital, Tokyo, Ota-ku
  - Sekino Hospital, Tokyo, Toshima-ku
  - Minami Wakayama Medical Center, Wakayama, Tanabe
  - Kanmon Medical Center, Yamaguchi, Shimonoseki
- Mexico (15):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Centro de Investigacion Biomedica y Farmaceutica, S.C., Distrito Federal
  - Unidad de Investigacion Clinica Cardiometabolica de Occident, Guadalajara
  - Diseño y Planeación en Investigación Médica SC, Guadalajara
  - Cardiologia Clinica e Intervencionista, Guadalajara
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Centro de Investigación Clinica Acelerada, S.C., México
  - CEDOPEC-Ctro Esp en Diab, Obesidad y Prev de Enf Cardiovasc, México
  - Instituto Cardiovascular de Monclova, S de RL de CV, Monclova
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Nuevo León
  - Centro Integral Medico SJR S.C., San Juan del Río
  - Cardioarritmias e Investigación S.C, San Luis Potosí City
  - Centro de Investigacion Cardiovascular y Metabolica, Tijuana
  - Centro de Investigacion Medica Alberto Bazzoni S.A. de C.V., Torreón
  - Hospital Dr Angel Leano, Zapopan
- Netherlands (23):
  - Ziekenhuisgroep Twente locatie Almelo, Almelo
  - BovenIJ Ziekenhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Locatie West, Amsterdam
  - Amsterdam UMC Locatie VUMC, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Rode Kruis Ziekenhuis Beverwijk, Beverwijk
  - Tergooiziekenhuizen locatie Blaricum, Blaricum
  - Amphia Ziekenhuis, Breda
  - Ziekenhuis Gelderse Vallei, Ede
  - Catharina Ziekenhuis, Eindhoven
  - Universitair Medisch Centrum Groningen, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Vasculair Onderzoek Centrum, Hoorn
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Diaconessenhuis Meppel, Meppel
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Radboud Universitair Medisch Centrum, Nijmegen
  - HMC Bronovo, The Hague
  - Ziekenhuis Bernhoven Uden, Uden
  - Vie Curi Medisch Centrum, Venlo
  - De Heel - Zaans Medisch Centrum, Zaandam
  - Gelre Ziekenhuis Zutphen, Zutphen
- Poland (33):
  - KLIMED Marek Klimkiewicz, Bialystok
  - Univ. Clinic Hosp, Bialystok, Bialystok
  - American Heart of Poland Sp. z o.o., Bielsko-Biala
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - Polsko-Amerykanskie Kliniki Serca, Chorzów
  - American Heart of Poland Sp. z o.o., Dąbrowa Górnicza
  - Poradnia Kardiologiczna Jaroslaw Jurowiecki, Gdansk
  - University Clinical Center, Gdansk, Gdansk
  - Indywidualna Specjalistyczna Praktyka Lekarska, Gdynia
  - Saint Wincenty a Paulo Hosp., Cardiology Dept., Gdynia, Gdynia
  - Szpital Zakonu Bonifratow Sp. z o.o., Katowice
  - Specialistic Cardiology&Hypertension Out-patient Clin,Kielce, Kielce
  - Leszek Bryniarski Specialized Medical Cabinet, Krakow
  - Krakow Specialistic Hospital of John Paul II, Krakow
  - SANTA FAMILIA Centrum Badan, Profilaktyki i Leczenia, Lodz
  - Nzoz Salus, Lodz
  - Individual Specialized Practice, Lodz
  - Lowickie Cardiology Center, Lowicz
  - American Heart of Poland Sp. z o.o., Nysa
  - Medicome Sp. z o.o., Oświęcim
  - Specialized Practice Dr. Janusz Spyra, Ruda Śląska
  - Centrum Medyczne Medyk, Rzeszów
  - Lukmed Lukasz Wozniak, Siedlce
  - Clinmedica Research Omc sp. z o.o. sp.k., Skierniewice, Skierniewice
  - KO-MED Centra Kliniczne Staszow, Staszów
  - The Provincial Polyclinical Hospital in Torun, Torun
  - American Heart of Poland Sp. z o.o., Tychy
  - American Heart of Poland Sp. z o.o., Ustroń
  - Central Hospital of Medical Academy, Warsaw, Warsaw
  - McM Polimedica, Warsaw
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
  - Zgierskie Center of Cardiology MED-PRO, Zgierz
  - Specialist Hospital J. Dietla NZOZ Specialized Clinic "Gemini", Żychlin
- South Korea (12):
  - Dong-A University Hospital, Busan
  - Inje University Busan Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Bundang Hospital, Sungnam
  - Wonju Severance Christian Hosp, Wŏnju
- Spain (12):
  - Hospital Quiron. I.C.U., Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Complejo Hospitalario Universitario de Orense, Ourense
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (9):
  - Barnet General Hospital, Barnet
  - University Hospital of Wales, Cardiff
  - Park & St Francis Surgery, Eastleigh
  - Wycombe General Hospital, High Wycombe
  - Glenfield Hospital, Leicester
  - St Bartholomew's Hospital, London
  - Luton and Dunstable University Hospital, Luton
  - St Mary's Hospital, Newport
  - Morriston Hospital, Swansea

REFERENCES:
- [Derived] Packer M, Ferreira JP, Butler J, Filippatos G, Januzzi JL Jr, Gonzalez Maldonado S, Panova-Noeva M, Pocock SJ, Prochaska JH, Saadati M, Sattar N, Sumin M, Anker SD, Zannad F. Reaffirmation of Mechanistic Proteomic Signatures Accompanying SGLT2 Inhibition in Patients With Heart Failure: A Validation Cohort of the EMPEROR Program. J Am Coll Cardiol. 2024 Nov 12;84(20):1979-1994. doi: 10.1016/j.jacc.2024.07.013. Epub 2024 Aug 31. PMID 39217550
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Ferreira JP, Packer M, Sattar N, Butler J, Pocock SJ, Anker SD, Maldonado SG, Panova-Noeva M, Sumin M, Masson S, Zannad F, Januzzi JL. Carbohydrate antigen 125 concentrations across the ejection fraction spectrum in chronic heart failure: The EMPEROR programme. Eur J Heart Fail. 2024 Apr;26(4):788-802. doi: 10.1002/ejhf.3166. Epub 2024 Mar 4. PMID 38439582
- [Derived] Zannad F, Macari S. Drug treatment with empagliflozin lowered risk for hospitalization in people with heart failure with reduced ejection fraction: plain language summary of the EMPEROR-Reduced study. Future Cardiol. 2023 Oct;19(13):625-630. doi: 10.2217/fca-2023-0090. Epub 2023 Nov 9. PMID 37942680
- [Derived] Dhingra NK, Verma S, Butler J, Anker SD, Ferreira JP, Filippatos G, Januzzi JL, Lam CSP, Sattar N, Zaremba-Pechmann L, Bohm M, Nordaby M, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Reduced Trial Committees and Investigators. Efficacy and Safety of Empagliflozin According to Background Diuretic Use in HFrEF: Post-Hoc Analysis of EMPEROR-Reduced. JACC Heart Fail. 2024 Jan;12(1):35-46. doi: 10.1016/j.jchf.2023.06.036. Epub 2023 Sep 13. PMID 37715769
- [Derived] Packer M, Butler J, Zeller C, Pocock SJ, Brueckmann M, Ferreira JP, Filippatos G, Usman MS, Zannad F, Anker SD. Blinded Withdrawal of Long-Term Randomized Treatment With Empagliflozin or Placebo in Patients With Heart Failure. Circulation. 2023 Sep 26;148(13):1011-1022. doi: 10.1161/CIRCULATIONAHA.123.065748. Epub 2023 Aug 24. PMID 37621153
- [Derived] Carson P, Teerlink JR, Komajda M, Anand I, Anker SD, Butler J, Doehner W, Ferreira JP, Filippatos G, Haass M, Miller A, Pehrson S, Pocock SJ, Schnaidt S, Schnee JM, Zannad F, Packer M. Comparison of Investigator-Reported and Centrally Adjudicated Heart Failure Outcomes in the EMPEROR-Reduced Trial. JACC Heart Fail. 2023 Apr;11(4):407-417. doi: 10.1016/j.jchf.2022.11.017. Epub 2023 Feb 1. PMID 36881400
- [Derived] Khan MS, Butler J, Anker SD, Filippatos G, Ferreira JP, Pocock SJ, Januzzi JL, Pina IL, Bohm M, Ponikowski P, Verma S, Brueckmann M, Vedin O, Zeller C, Zannad F, Packer M. Impact of Empagliflozin in Heart Failure With Reduced Ejection Fraction in Patients With Ischemic Versus Nonischemic Cause. J Am Heart Assoc. 2023 Jan 3;12(1):e027652. doi: 10.1161/JAHA.122.027652. Epub 2022 Dec 24. PMID 36565199
- [Derived] Ferreira JP, Zannad F, Butler J, Filippatos G, Pocock SJ, Brueckmann M, Steubl D, Schueler E, Anker SD, Packer M. Association of Empagliflozin Treatment With Albuminuria Levels in Patients With Heart Failure: A Secondary Analysis of EMPEROR-Pooled. JAMA Cardiol. 2022 Nov 1;7(11):1148-1159. doi: 10.1001/jamacardio.2022.2924. PMID 36129693
- [Derived] Zannad F, Ferreira JP, Butler J, Filippatos G, Januzzi JL, Sumin M, Zwick M, Saadati M, Pocock SJ, Sattar N, Anker SD, Packer M. Effect of empagliflozin on circulating proteomics in heart failure: mechanistic insights into the EMPEROR programme. Eur Heart J. 2022 Dec 21;43(48):4991-5002. doi: 10.1093/eurheartj/ehac495. PMID 36017745
- [Derived] Zannad F, Ferreira JP, Gregson J, Kraus BJ, Mattheus M, Hauske SJ, Butler J, Filippatos G, Wanner C, Anker SD, Pocock SJ, Packer M; EMPEROR-Reduced Trial Committees and Investigators. Early changes in estimated glomerular filtration rate post-initiation of empagliflozin in EMPEROR-Reduced. Eur J Heart Fail. 2022 Oct;24(10):1829-1839. doi: 10.1002/ejhf.2578. Epub 2022 Jul 7. PMID 35711093
- [Derived] Ferreira JP, Zannad F, Butler J, Filipattos G, Ritter I, Schuler E, Kraus BJ, Pocock SJ, Anker SD, Packer M. Empagliflozin and serum potassium in heart failure: an analysis from EMPEROR-Pooled. Eur Heart J. 2022 Aug 14;43(31):2984-2993. doi: 10.1093/eurheartj/ehac306. PMID 35687107
- [Derived] Ferreira JP, Butler J, Zannad F, Filippatos G, Schueler E, Steubl D, Zeller C, Januzzi JL, Pocock S, Packer M, Anker SD. Mineralocorticoid Receptor Antagonists and Empagliflozin in Patients With Heart Failure and Preserved Ejection Fraction. J Am Coll Cardiol. 2022 Mar 29;79(12):1129-1137. doi: 10.1016/j.jacc.2022.01.029. PMID 35331406
- [Derived] Ferreira JP, Anker SD, Butler J, Filippatos G, Iwata T, Salsali A, Zeller C, Pocock SJ, Zannad F, Packer M. Impact of anaemia and the effect of empagliflozin in heart failure with reduced ejection fraction: findings from EMPEROR-Reduced. Eur J Heart Fail. 2022 Apr;24(4):708-715. doi: 10.1002/ejhf.2409. Epub 2022 Jan 9. PMID 34957660
- [Derived] Verma S, Dhingra NK, Butler J, Anker SD, Ferreira JP, Filippatos G, Januzzi JL, Lam CSP, Sattar N, Peil B, Nordaby M, Brueckmann M, Pocock SJ, Zannad F, Packer M; EMPEROR-Reduced trial committees and investigators. Empagliflozin in the treatment of heart failure with reduced ejection fraction in addition to background therapies and therapeutic combinations (EMPEROR-Reduced): a post-hoc analysis of a randomised, double-blind trial. Lancet Diabetes Endocrinol. 2022 Jan;10(1):35-45. doi: 10.1016/S2213-8587(21)00292-8. Epub 2021 Nov 30. PMID 34861154
- [Derived] Ryden L, Ferrannini G. Is the impact of add on heart failure therapy influenced by background therapy? Lancet Diabetes Endocrinol. 2022 Jan;10(1):3-5. doi: 10.1016/S2213-8587(21)00311-9. Epub 2021 Nov 30. No abstract available. PMID 34861151
- [Derived] Bohm M, Anker SD, Butler J, Filippatos G, Ferreira JP, Pocock SJ, Mahfoud F, Brueckmann M, Jamal W, Ofstad AP, Schuler E, Ponikowski P, Wanner C, Zannad F, Packer M; EMPEROR-Reduced Trial Committees and Investigators. Empagliflozin Improves Cardiovascular and Renal Outcomes in Heart Failure Irrespective of Systolic Blood Pressure. J Am Coll Cardiol. 2021 Sep 28;78(13):1337-1348. doi: 10.1016/j.jacc.2021.07.049. PMID 34556320
- [Derived] Januzzi JL Jr, Zannad F, Anker SD, Butler J, Filippatos G, Pocock SJ, Ferreira JP, Sattar N, Verma S, Vedin O, Schnee J, Iwata T, Cotton D, Packer M; EMPEROR-Reduced Trial Committees and Investigators. Prognostic Importance of NT-proBNP and Effect of Empagliflozin in the EMPEROR-Reduced Trial. J Am Coll Cardiol. 2021 Sep 28;78(13):1321-1332. doi: 10.1016/j.jacc.2021.07.046. PMID 34556318
- [Derived] Packer M, Butler J, Zannad F, Filippatos G, Ferreira JP, Pocock SJ, Carson P, Anand I, Doehner W, Haass M, Komajda M, Miller A, Pehrson S, Teerlink JR, Schnaidt S, Zeller C, Schnee JM, Anker SD. Effect of Empagliflozin on Worsening Heart Failure Events in Patients With Heart Failure and Preserved Ejection Fraction: EMPEROR-Preserved Trial. Circulation. 2021 Oct 19;144(16):1284-1294. doi: 10.1161/CIRCULATIONAHA.121.056824. Epub 2021 Aug 29. PMID 34459213
- [Derived] Pocock SJ, Ferreira JP, Gregson J, Anker SD, Butler J, Filippatos G, Gollop ND, Iwata T, Brueckmann M, Januzzi JL, Voors AA, Zannad F, Packer M. Novel biomarker-driven prognostic models to predict morbidity and mortality in chronic heart failure: the EMPEROR-Reduced trial. Eur Heart J. 2021 Nov 14;42(43):4455-4464. doi: 10.1093/eurheartj/ehab579. PMID 34423361
- [Derived] Lam CSP, Ferreira JP, Pfarr E, Sim D, Tsutsui H, Anker SD, Butler J, Filippatos G, Pocock SJ, Sattar N, Verma S, Brueckmann M, Schnee J, Cotton D, Zannad F, Packer M. Regional and ethnic influences on the response to empagliflozin in patients with heart failure and a reduced ejection fraction: the EMPEROR-Reduced trial. Eur Heart J. 2021 Nov 14;42(43):4442-4451. doi: 10.1093/eurheartj/ehab360. PMID 34184057
- [Derived] Ferreira JP, Zannad F, Pocock SJ, Anker SD, Butler J, Filippatos G, Brueckmann M, Jamal W, Steubl D, Schueler E, Packer M. Interplay of Mineralocorticoid Receptor Antagonists and Empagliflozin in Heart Failure: EMPEROR-Reduced. J Am Coll Cardiol. 2021 Mar 23;77(11):1397-1407. doi: 10.1016/j.jacc.2021.01.044. PMID 33736821
- [Derived] Packer M, Anker SD, Butler J, Filippatos G, Ferreira JP, Pocock SJ, Sattar N, Brueckmann M, Jamal W, Cotton D, Iwata T, Zannad F; EMPEROR-Reduced Trial Committees and Investigators. Empagliflozin in Patients With Heart Failure, Reduced Ejection Fraction, and Volume Overload: EMPEROR-Reduced Trial. J Am Coll Cardiol. 2021 Mar 23;77(11):1381-1392. doi: 10.1016/j.jacc.2021.01.033. PMID 33736819
- [Derived] Butler J, Anker SD, Filippatos G, Khan MS, Ferreira JP, Pocock SJ, Giannetti N, Januzzi JL, Pina IL, Lam CSP, Ponikowski P, Sattar N, Verma S, Brueckmann M, Jamal W, Vedin O, Peil B, Zeller C, Zannad F, Packer M; EMPEROR-Reduced Trial Committees and Investigators. Empagliflozin and health-related quality of life outcomes in patients with heart failure with reduced ejection fraction: the EMPEROR-Reduced trial. Eur Heart J. 2021 Mar 31;42(13):1203-1212. doi: 10.1093/eurheartj/ehaa1007. PMID 33420498
- [Derived] Anker SD, Butler J, Filippatos G, Khan MS, Marx N, Lam CSP, Schnaidt S, Ofstad AP, Brueckmann M, Jamal W, Bocchi EA, Ponikowski P, Perrone SV, Januzzi JL, Verma S, Bohm M, Ferreira JP, Pocock SJ, Zannad F, Packer M. Effect of Empagliflozin on Cardiovascular and Renal Outcomes in Patients With Heart Failure by Baseline Diabetes Status: Results From the EMPEROR-Reduced Trial. Circulation. 2021 Jan 26;143(4):337-349. doi: 10.1161/CIRCULATIONAHA.120.051824. Epub 2020 Nov 11. PMID 33175585
- [Derived] Zannad F, Ferreira JP, Pocock SJ, Zeller C, Anker SD, Butler J, Filippatos G, Hauske SJ, Brueckmann M, Pfarr E, Schnee J, Wanner C, Packer M. Cardiac and Kidney Benefits of Empagliflozin in Heart Failure Across the Spectrum of Kidney Function: Insights From EMPEROR-Reduced. Circulation. 2021 Jan 26;143(4):310-321. doi: 10.1161/CIRCULATIONAHA.120.051685. Epub 2020 Oct 23. PMID 33095032
- [Derived] Packer M, Anker SD, Butler J, Filippatos G, Ferreira JP, Pocock SJ, Carson P, Anand I, Doehner W, Haass M, Komajda M, Miller A, Pehrson S, Teerlink JR, Brueckmann M, Jamal W, Zeller C, Schnaidt S, Zannad F. Effect of Empagliflozin on the Clinical Stability of Patients With Heart Failure and a Reduced Ejection Fraction: The EMPEROR-Reduced Trial. Circulation. 2021 Jan 26;143(4):326-336. doi: 10.1161/CIRCULATIONAHA.120.051783. Epub 2020 Oct 21. PMID 33081531
- [Derived] Packer M, Anker SD, Butler J, Filippatos G, Pocock SJ, Carson P, Januzzi J, Verma S, Tsutsui H, Brueckmann M, Jamal W, Kimura K, Schnee J, Zeller C, Cotton D, Bocchi E, Bohm M, Choi DJ, Chopra V, Chuquiure E, Giannetti N, Janssens S, Zhang J, Gonzalez Juanatey JR, Kaul S, Brunner-La Rocca HP, Merkely B, Nicholls SJ, Perrone S, Pina I, Ponikowski P, Sattar N, Senni M, Seronde MF, Spinar J, Squire I, Taddei S, Wanner C, Zannad F; EMPEROR-Reduced Trial Investigators. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. N Engl J Med. 2020 Oct 8;383(15):1413-1424. doi: 10.1056/NEJMoa2022190. Epub 2020 Aug 28. PMID 32865377
- [Derived] Nassif ME, Kosiborod M. Effects of sodium glucose cotransporter type 2 inhibitors on heart failure. Diabetes Obes Metab. 2019 Apr;21 Suppl 2:19-23. doi: 10.1111/dom.13678. PMID 31081589
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomised, double-blind trial to demonstrate superiority of empagliflozin versus placebo, in patients with chronic Heart Failure with reduced Ejection Fraction (HFrEF).
Pre-assignment Details: Patients were included in the trial after they had signed the informed consent form (ICF). All patients who met the all inclusion and none of the exclusion criteria during screening and at the randomisation approximately 1 to 4 weeks later were randomised to empagliflozin or placebo in a 1:1 ratio.
Groups:
- Placebo: 1 film-coated tablet of matching placebo was administered orally once daily.
- 10 mg Empagliflozin: Film-coated tablet of 10 milligram (mg) Empagliflozin was administered orally once daily.
Period: Discontinuation From Treatment
Arm/Group | Placebo | 10 mg Empagliflozin
Started (Randomized) | 1867 | 1863
Treated | 1863 | 1863
Completed (Completed treatment) | 1352 | 1381
Not Completed | 515 | 482
Not completed — Withdrawal by Subject | 124 | 92
Not completed — Lost to Follow-up | 11 | 17
Not completed — Protocol Violation | 6 | 5
Not completed — Not treated | 4 | 0
Not completed — Adverse Event | 343 | 337
Not completed — Reason Unknown | 0 | 1
Not completed — Personal Reasons | 1 | 1
Not completed — Unblinded medication | 1 | 0
Not completed — Patient received Empagliflozin for Diabetes | 1 | 1
Not completed — Principle Investigator Decision | 2 | 0
Not completed — Other medical condition (no Adverse Event) | 2 | 4
Not completed — Patient moved away/being abroad | 4 | 3
Not completed — Unable to continue treatment | 4 | 1
Not completed — Not attending study visit | 3 | 10
Not completed — Due to Covid-19 Pandemic | 1 | 4
Not completed — Patient decision to stop/interrupt medication | 8 | 6
Period: Discontinuation From Trial
Arm/Group | Placebo | 10 mg Empagliflozin
Started (Randomized) | 1867 | 1863
Treated | 1863 | 1863
Completed | 1847 | 1841
Not Completed | 20 | 22
Not completed — Lost to follow-up to primary endpoint | 9 | 9
Not completed — Limited follow-up agreed | 2 | 2
Not completed — Withdrawal by Subject | 9 | 11

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): All randomised patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Empagliflozin | Total
Number analyzed (Participants) | 1867 | 1863 | 3730
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (11.2) | 67.2 (10.8) | 66.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 456 | 437 | 893
  Male | 1411 | 1426 | 2837
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 613 | 616 | 1229
  Not Hispanic or Latino | 1178 | 1164 | 2342
  Unknown or Not Reported | 76 | 83 | 159
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 24 | 15 | 39
  Asian | 335 | 337 | 672
  Native Hawaiian or Other Pacific Islander | 6 | 8 | 14
  Black or African American | 134 | 123 | 257
  White | 1304 | 1325 | 2629
  More than one race | 33 | 28 | 61
  Unknown or Not Reported | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Time to the First Event of Adjudicated Cardiovascular (CV) Death or Adjudicated Hospitalisation for Heart Failure (HHF)
Description: Time to the first event of adjudicated cardiovascular (CV) death or adjudicated hospitalisation for heart failure (HHF). The incidence rate per 100 patient years (100 * number of patients with event /time at risk [years]) is presented. With time at risk [year] calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
  Unit of Measure: Patients with events per 100 patient-years (pt-yrs) at risk.
Time Frame: From randomisation until completion of the planned treatment period, up to 1040 days.
Population: Randomised Set: All randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with events/ 100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1867 | 1863
Patients with events/ 100 pt-yrs at risk | 21.00 [19.13 to 22.96] | 15.77 [14.19 to 17.44]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Model with terms for age, baseline eGFR (CKD-EPK)cr, region, baseline diabetes status, sex, baseline LVEF, and treatment. alpha = 0.0496 (resulting from interim analysis) eGFR (CKP-EPI)cr: Glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement LVEF: Left ventricular ejection fraction; Test type: Superiority — H0: There is no difference between the effect of placebo and the effect of empagliflozin; p < 0.0001, Regression, Cox; Hazard Ratio (HR) = 0.75, 95.04% CI 2-sided [0.65 to 0.86] — Comparison vs. Placebo [T/P]

2. Secondary Outcome: Occurrence of Adjudicated Hospitalisation for Heart Failure (HHF) (First and Recurrent)
Description: Reported is the total number of HHF events (first and recurrent) which occurred.
  All data up to the end of the planned treatment period (including the data after the end of treatment for patients not completing the treatment period as planned) from all randomised patients was used.
Time Frame: From randomisation until completion of the planned treatment phase, up to 1040 days.
Population: Randomised Set (RS): All randomised patients.
Measure: Number; unit: HHF events
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1867 | 1863
HHF events | 553 | 388
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Model accounts for dependence between recurrent HHF and cardiovascular death, with terms for age, baseline eGFR (CKD-EPK)cr, region, baseline diabetes status, sex, baseline LVEF, and treatment. eGFR (CKP-EPI)cr: Glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement LVEF: Left ventricular ejection fraction; Test type: Superiority — H0: There is no difference between the effect of placebo and the effect of empagliflozin; p = 0.0003, Joint frailty model; Hazard Ratio (HR) = 0.70, 95.04% CI 2-sided [0.58 to 0.85] — HR vs placebo of recurrent HFF

3. Secondary Outcome: eGFR (CKD-EPI) cr Slope of Change From Baseline
Description: Glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement (eGFR (CKD-EPI)cr) [mL/min/1.73m2] slope of change from baseline.
  Available on-treatment change-from-baseline data were to be used. Patients without on-treatment data after randomisation were not to be included in this analysis. Slope represents the long term effect on eGFR.
  Timepoints after baseline were included in calculation of slope of change from baseline. Descriptive statistic (mean(standard error)) is reported.
Time Frame: Assessed at baseline, week 4, 12, 32, 52, 76, 100, 124, 148 and at end of treatment (EOT), up to 1040 days.
Population: Treated Set (TS): All patients treated with at least one dose of the study medication and at least one on-treatment measurement of eGFR.
Measure: Mean (Standard Error); unit: Milliliter/minute/1.73 meters squared
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1792 | 1799
Milliliter/minute/1.73 meters squared | -2.278 (0.229) | -0.546 (0.227)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Random coefficient model allowing for random intercept and random slope per patient, with the same factors used for the primary endpoint (age, baseline eGFR (CKD-EPK)cr, region, baseline diabetes status, sex, baseline LVEF, and treatment) and additional factors "time", "treatment-by-time interaction", and "baseline eGFR (CKD-EPI)cr-by-time interaction". Only "on-treatment" data from treated patients were used. alpha=0.001; Test type: Superiority — H0: There is no difference between the effect of placebo and the effect of empagliflozin; p < 0.0001, Random intercept random coef. model; Treatment by time interaction = 1.733, 99.9% CI 2-sided [0.669 to 2.796] — Empa vs Placebo slope [/year]

4. Secondary Outcome: Time to First Event in Composite Renal Endpoint: Chronic Dialysis, Renal Transplant or Sustained Reduction of eGFR(CKD-EPI)cr
Description: Time to the first event in the composite renal endpoint: chronic dialysis (with a frequency of twice per week or more for at least 90 days), renal transplant, or sustained reduction in Glomerular filtration rate estimated by the chronic kidney disease epidemiology collaboration formula with serum creatinine measurement (eGFR (CKD-EPI)cr).
  The incidence rate per 100 patient years (100 * number of patients with event /time at risk [years]) is presented. With time at risk [year] calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
  Unit of Measure: Patients with events per 100 patient-years (pt-yrs) at risk.
Time Frame: From randomisation until completion of the planned treatment period, up to 1040 days.
Population: Randomised Set: All randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with events/ 100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1867 | 1863
Patients with events/ 100 pt-yrs at risk | 3.07 [2.33 to 3.91] | 1.56 [1.06 to 2.17]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.0019, Regression, Cox; Cox regression model with terms for age, baseline eGFR (CKD-EPK)cr, region, baseline diabetes status, sex, baseline LVEF, and treatment; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.32 to 0.77] — Comparison vs. Placebo

5. Secondary Outcome: Time to First Adjudicated Hospitalisation for Heart Failure (HHF)
Description: Time to first adjudicated Hospitalisation for Heart Failure (HHF). The incidence rate per 100 patient years (100 * number of patients with event /time at risk [years]) is presented. With time at risk [year] calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25. Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
  Unit of Measure: Patients with events per 100 patient-years (pt-yrs) at risk.
Time Frame: From randomisation until completion of the planned treatment period, up to 1040 days.
Population: Randomised Set (RS): All randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with events/ 100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1867 | 1863
Patients with events/ 100 pt-yrs at risk | 15.55 [13.94 to 17.24] | 10.75 [9.45 to 12.13]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p < 0.0001, Regression, Cox; [statistical method as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.59 to 0.81] — Comparison vs Placebo

6. Secondary Outcome: Time to Adjudicated Cardiovascular (CV) Death
Description: Time to adjudicated CV (Cardiovascular) death. The incidence rate (patients with events per 100 person years at risk) is reported.
  The incidence rate per 100 patient years (100 * number of patients with event /time at risk [years]) is presented. With time at risk [year] calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
  Unit of Measure: Patients with events per 100 patient-years (pt-yrs) at risk.
Time Frame: From randomisation until completion of the planned treatment period, up to 1040 days.
Population: Randomised Set: All randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with events/ 100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1867 | 1863
Patients with events/ 100 pt-yrs at risk | 8.13 [7.05 to 9.29] | 7.55 [6.51 to 8.67]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.4133, Regression, Cox; Model with terms for age, baseline eGFR (CKD-EPI), region, baseline diabetes status, sex, baseline LVEF and treatment; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.75 to 1.12] — Comparison vs. Placebo

7. Secondary Outcome: Time to All-cause Mortality
Description: Time to all-cause mortality. The incidence rate (patients with events per 100 person years at risk) is reported.
  The incidence rate per 100 patient years (100 * number of patients with event /time at risk [years]) is presented. With time at risk [year] calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
  Unit of Measure: Patients with events per 100 patient-years (pt-yrs) at risk.
Time Frame: From randomisation until completion of the planned treatment period, up to 1040 days.
Population: Randomised Set: All randomised patients.
Measure: Number (95% Confidence Interval); unit: Patients with events/ 100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1867 | 1863
Patients with events/ 100 pt-yrs at risk | 10.71 [9.46 to 12.04] | 10.06 [8.85 to 11.34]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.3536, Regression, Cox; Cox regression model with terms for age, baseline eGFR (CKD-EPI), region, baseline diabetes status, sex, baseline LVEF and treatment; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.77 to 1.10] — Comparison vs. placebo

8. Secondary Outcome: Time to Onset of Diabetes Mellitus (DM)
Description: Time to onset of DM (Glycated haemoglobin (HbA1c) ≥6.5% or as diagnosed by the investigator) in patients with pre-DM (no history of DM and no HbA1c ≥6.5% before treatment, and a pre-treatment HbA1c value of 5.7 to <6.5%). The incidence rate (patients with events per 100 person years at risk) is reported.
  The incidence rate per 100 patient years (100 * number of patients with event /time at risk [years]) is presented. With time at risk [year] calculated as: Sum of time at risk [days] over all patients in a treatment group / 365.25.
  Patients without a specific endpoint event were censored at the last date the patient was known to be free of the event or at the end of the planned treatment period, whichever was earlier.
  Unit of Measure: Patients with events per 100 patient-years (pt-yrs) at risk.
Time Frame: From randomisation until completion of the planned treatment period, up to 1040 days.
Population: Patients in the randomised set with pre-DM.
Measure: Number (95% Confidence Interval); unit: Patients with events/ 100 pt-yrs at risk
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 636 | 632
Patients with events/ 100 pt-yrs at risk | 10.62 [8.42 to 13.07] | 9.31 [7.27 to 11.60]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Test type: Other; p = 0.3576, Regression, Cox; Cox regression model with terms for age, baseline eGFR (CDK-EPI), region, sex, baseline LVEF and treatment; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.62 to 1.19] — Comparison vs. placebo

9. Secondary Outcome: Change From Baseline in KCCQ (Kansas City Cardiomyopathy Questionnaire) Clinical Summary Score at Week 52
Description: Change from baseline in KCCQ (Kansas City cardiomyopathy questionnaire) clinical summary score at Week 52. The KCCQ is a 23-item self-administered questionnaire designed to evaluate physical limitations, symptoms (frequency, severity, and changes over time), social limitations, selfefficacy, and quality of life in patients with Heart Failure. The KCCQ-clinical summary score comprises the following domains: Symptom frequency, symptom burden and physical limitation. The score is calculated by summing domain responses and then transforming scores to a 0-100 unit scale with higher scores indicating better health status.
  For patients who died, a worst score (score of 0) is imputed at all subsequent scheduled visits after the date of death.
  Standard error is adjusted standard error. Change from baseline in KCCQ-score at week 52 was modeled using a MMRM with visit (week 12, 32 and 52) as repeated measures, adjusted mean (standard error) at week 52 is reported.
Time Frame: Assessed at baseline, week 12, week 32 and week 52.
Population: Patients in the randomized set (RS) with available data for this endpoint, including values obtained on treatment or post-treatment.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1395 | 1401
Score on a scale | -3.36 (0.69) | -1.30 (0.69)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Mixed model with age, baseline eGFR (CKD-EPI) as linear covariate(s) and region, baseline diabetes status, sex, baseline LVEF, week reachable, treatment by visit interaction, baseline KCCQ - Clinical Summary Score by Visit interaction as fixed effects. An unstructured covariance structure has been used; Test type: Other; p = 0.0340, Mixed Model; Mixed model for repeated measures (MMRM); Difference of adjusted means = 2.06, 95% CI 2-sided [0.16 to 3.96], Standard Error of Mean 0.97 — Comparison vs. placebo

10. Secondary Outcome: Number of All-cause Hospitalizations (First and Recurrent)
Description: Number of all-cause hospitalizations (first and recurrent).
Time Frame: From randomisation until completion of the planned treatment phase, up to 1040 days.
Population: Randomised Set: All randomised patients.
Measure: Number; unit: Hospitalizations for any cause
Arm/Group | Placebo | 10 mg Empagliflozin
Number analyzed (Participants) | 1867 | 1863
Hospitalizations for any cause | 1570 | 1364
Statistical Analysis 1: Comparison: Placebo vs 10 mg Empagliflozin; Joint frailty model with terms for age, baseline eGFR (CDK-EPI), region, sex, baseline diabetes status and baseline LVEF. Model accounts for dependence between recurrent all-cause hospitalizations and all-cause mortality; Test type: Other; p = 0.0065, Joint frailty model; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.75 to 0.95] — Comparison vs. placebo

ADVERSE EVENTS:
Time Frame: From first intake of study medication until end of planned treatment period + 7 days (Residual Effect Period), up to 1047 days.
Description: [All-Cause Mortality]: Randomised Set: All randomised patients. [Serious Adverse Events and Other Adverse Events]: Treated Set: All patients treated with at least one dose of study drug.
Arm/Group | Placebo | 10 mg Empagliflozin
All-Cause Mortality (participants affected / at risk) | 266/1867 | 249/1863
Serious Adverse Events (participants affected / at risk) | 896/1863 | 772/1863
Other Adverse Events (participants affected / at risk) | 369/1863 | 328/1863
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1863) | 10 mg Empagliflozin (N=1863)
Anaemia (Blood and lymphatic system disorders) | 6 | 10
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Splenic haematoma (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 0
Acute left ventricular failure (Cardiac disorders) | 5 | 7
Acute myocardial infarction (Cardiac disorders) | 18 | 24
Angina pectoris (Cardiac disorders) | 10 | 6
Angina unstable (Cardiac disorders) | 9 | 11
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 44 | 24
Atrial flutter (Cardiac disorders) | 11 | 3
Atrial tachycardia (Cardiac disorders) | 2 | 4
Atrial thrombosis (Cardiac disorders) | 2 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 4
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 4 | 0
Bundle branch block left (Cardiac disorders) | 1 | 1
Cardiac aneurysm (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 10 | 9
Cardiac asthma (Cardiac disorders) | 0 | 2
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 444 | 332
Cardiac failure acute (Cardiac disorders) | 29 | 19
Cardiac failure chronic (Cardiac disorders) | 32 | 18
Cardiac failure congestive (Cardiac disorders) | 41 | 26
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 2 | 5
Cardio-respiratory arrest (Cardiac disorders) | 4 | 1
Cardiogenic shock (Cardiac disorders) | 11 | 8
Cardiomegaly (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Cardiorenal syndrome (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 6 | 1
Coronary artery disease (Cardiac disorders) | 16 | 2
Coronary artery occlusion (Cardiac disorders) | 3 | 3
Coronary artery stenosis (Cardiac disorders) | 2 | 3
Coronary ostial stenosis (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 2 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Left ventricular failure (Cardiac disorders) | 3 | 3
Low cardiac output syndrome (Cardiac disorders) | 1 | 2
Mitral valve incompetence (Cardiac disorders) | 5 | 4
Myocardial infarction (Cardiac disorders) | 16 | 16
Myocardial ischaemia (Cardiac disorders) | 1 | 3
Palpitations (Cardiac disorders) | 1 | 0
Paroxysmal atrioventricular block (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 6 | 2
Torsade de pointes (Cardiac disorders) | 0 | 1
Trifascicular block (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 5 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 2
Ventricular fibrillation (Cardiac disorders) | 8 | 10
Ventricular flutter (Cardiac disorders) | 1 | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 37 | 55
Dermoid cyst (Congenital, familial and genetic disorders) | 2 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 1
Type IV hyperlipidaemia (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Mixed deafness (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Cushing's syndrome (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 2 | 3
Hypothyroidism (Endocrine disorders) | 2 | 0
Cataract (Eye disorders) | 3 | 5
Cataract cortical (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 5 | 3
Macular degeneration (Eye disorders) | 1 | 0
Open angle glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 3
Retinal tear (Eye disorders) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric mucosa erythema (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 8
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 7
Intestinal ischaemia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Intussusception (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 1 | 0
Cardiac death (General disorders) | 8 | 4
Chest pain (General disorders) | 2 | 2
Death (General disorders) | 27 | 20
Discomfort (General disorders) | 1 | 0
Euthanasia (General disorders) | 0 | 1
Foreign body reaction (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Implant site haematoma (General disorders) | 1 | 0
Medical device site haematoma (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 7 | 5
Oedema due to cardiac disease (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 3
Pyrexia (General disorders) | 1 | 1
Stent-graft endoleak (General disorders) | 2 | 0
Sudden cardiac death (General disorders) | 10 | 8
Sudden death (General disorders) | 5 | 5
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Vascular device occlusion (General disorders) | 1 | 0
Vessel puncture site phlebitis (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Cardiac cirrhosis (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 5 | 2
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 5 | 3
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0
Heart transplant rejection (Immune system disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 3 | 3
Appendicitis perforated (Infections and infestations) | 0 | 2
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 5 | 5
Bullous erysipelas (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 3 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 8
Clostridium difficile infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 2
Diabetic foot infection (Infections and infestations) | 0 | 3
Disseminated tuberculosis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Encephalitis viral (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 3 | 2
Erysipelas (Infections and infestations) | 3 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Eye abscess (Infections and infestations) | 1 | 0
Fournier's gangrene (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 4
Gastritis viral (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 9 | 4
Gastrointestinal infection (Infections and infestations) | 2 | 1
Haemorrhagic fever (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Human anaplasmosis (Infections and infestations) | 0 | 1
Implant site infection (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Infective spondylitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 5 | 4
Intervertebral discitis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Medical device site infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 2
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 2
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 62 | 53
Pneumonia bacterial (Infections and infestations) | 3 | 1
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 2 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 2
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 2 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 8 | 8
Septic encephalopathy (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 5 | 9
Sinobronchitis (Infections and infestations) | 1 | 0
Spinal cord abscess (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 10 | 14
Urosepsis (Infections and infestations) | 0 | 4
Vessel puncture site cellulitis (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 3 | 2
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 2
Bladder injury (Injury, poisoning and procedural complications) | 0 | 1
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Costal cartilage fracture (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 15
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 3 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 3
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Open globe injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1
Procedural shock (Injury, poisoning and procedural complications) | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 4
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 6
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Cardiac electrophysiologic study (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Endoscopic retrograde cholangiopancreatography (Investigations) | 1 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Diabetic complication (Metabolism and nutrition disorders) | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 7 | 2
Gout (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 4
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Bladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Cutaneous T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 6
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cerebral hypoperfusion (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 2 | 4
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 12 | 17
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 3 | 2
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hyperglycaemic seizure (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 20 | 19
Lacunar infarction (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 2
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 1 | 1
Postresuscitation encephalopathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 4
Seizure (Nervous system disorders) | 3 | 2
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 8 | 17
Transient ischaemic attack (Nervous system disorders) | 9 | 5
Uraemic encephalopathy (Nervous system disorders) | 1 | 0
Vascular dementia (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Device breakage (Product Issues) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Device failure (Product Issues) | 0 | 1
Device inappropriate shock delivery (Product Issues) | 0 | 1
Device lead damage (Product Issues) | 1 | 0
Device lead issue (Product Issues) | 0 | 2
Device malfunction (Product Issues) | 4 | 3
Device physical property issue (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 4 | 8
Delirium tremens (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Drug abuse (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 55 | 35
Azotaemia (Renal and urinary disorders) | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 6 | 3
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1
End stage renal disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 2
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 14 | 9
Renal impairment (Renal and urinary disorders) | 27 | 17
Renal infarct (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 3
Urethral stenosis (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 6
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 4
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 | 1
Cardioversion (Surgical and medical procedures) | 1 | 0
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 2 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Aortic intramural haematoma (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 2 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 5 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 4
Diabetic vascular disorder (Vascular disorders) | 1 | 0
Dry gangrene (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 2
Femoral artery embolism (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 4 | 6
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 13 | 14
Hypovolaemic shock (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1
Leriche syndrome (Vascular disorders) | 0 | 2
Lymphocele (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 4
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 7
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 4 | 5
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subclavian artery occlusion (Vascular disorders) | 1 | 1
Subclavian vein occlusion (Vascular disorders) | 1 | 0
Subgaleal haemorrhage (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Vascular insufficiency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1863) | 10 mg Empagliflozin (N=1863)
Nasopharyngitis (Infections and infestations) | 94 | 89
Hyperkalaemia (Metabolism and nutrition disorders) | 109 | 99
Hyperuricaemia (Metabolism and nutrition disorders) | 115 | 63
Hypotension (Vascular disorders) | 109 | 120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT03057977/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03057977/SAP_001.pdf